CLINICAL TRIAL: NCT00342511
Title: Pilots of Self-Collection Devices for HPV DNA Detection
Brief Title: Pilots of Self-Collection for HPV DNA Detection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906075; 06-C-N075
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-13

CONDITIONS: HPV
Keywords: Pap; Hybrid Capture 2; HSIL; Colposcopy; CIN; Specimen Collection

SUMMARY:
This study will evaluate a method of testing for human papillomavirus (HPV) DNA. For women who have had Pap test results that are abnormal, a new test can be done for HPV, that is, viruses that sometimes cause bumpy or flat warts. Such infections all usually disappear by themselves in 1 or 2 years if someone's Pap test shows a mild abnormality. But if the HPV does not go away, the infection can slowly lead to cancer of the cervix. Through this study, researchers will examine patients in conjunction with a colposcopy, that is, a diagnostic tool to determine the cause of abnormal Pap test results. The researchers hope to improve on the efficiency of detecting HPV and reducing the risk of cervical cancer.

Patients ages 21 and older who are not pregnant and who have not had a hysterectomy and who are attending a colposcopy clinic may be eligible for this study. This study will enroll 150 patients. Two pilot studies will be done: one at the Cleveland Clinic, with the use of the POI sampler (Preventive Oncology International ) and the other at the University of Arizona, with the use of the Fournier sampler.

In the study part that uses the POI sampler, patients will be recruited from the existing colposcopy schedule. For the Fournier sampler, patients will be recruited as they attend their scheduled colposcopy visit. During the procedure, the doctor will collect two (Cleveland Clinic) or three (University of Arizona) specimen from the patients while the patients are sitting. A speculum is not placed in the vagina at that time. Then the doctor will conduct a routine pelvic exam, with the use of a speculum, while the patients are lying down, and perform the colposcopy. One final specimen will be collected before the the colposcopic evaluation. Those three or four specimens will be used just for research purposes, and they make up the only part different from the regular colposcopy exam. The pelvic exams may sometimes be slightly uncomfortable, and patients may have temporary vaginal spotting of blood afterward. The collection of additional specimens may also cause slight discomfort.

The research specimens, which will not be labeled with information that directly identifies the patients, will be stored at a repository sponsored by NIH. Those specimens would be tested now or in the future.

Participants will be told about the results of their tests as part of the routine management of their abnormal Pap results. Women participating at the University of Arizona will receive $25 for the time they spend in the study. Benefits that patients receive from being part of this study include helping researchers to discover new ways to prevent cervical cancer.

DETAILED DESCRIPTION:
Background:

Cytology screening programs have efficiently reduced cervical cancer incidence and mortality in the U.S. by > 75%. However, these programs rely on the insensitive Pap smear and, consequently, are inefficient and overly expensive. Therefore, the needs of undeserved populations are not well-served by the current cytology-based programs for cervical cancer screening. Based on the central role of oncogenic types of human papillomavirus (HPV) causing virtually all cases of cervical cancer, HPV DVA testing is already approved by the FDA as an adjunctive screening modality to cytology in this country and as a primary screening modality internationally. A validated screening program of HPV DNA testing of self-collected cervicovaginal specimens might provide more sensitive and wider coverage screening than cytology in the populations underserved by cytology-based (Papanicolaou [Pap] smear or liquid-based cytology) screening programs and therefore are at an elevated risk of cervical cancer. We are currently evaluating self-collection devices for optimal detection of HPV DNA, including one (POI sampler) designed by Jerry Belinson (Cleveland Clinic) and one (Fournier device) by Arthur Fournier (University of Miami).

Objective:

To compare HPV DNA detection in cervicovaginal specimens collected using newly developed self-collection devices, the POI sampler or the Fournier device, to HPV DNA detection in cervicovaginal specimens collected using a Darcon swab and HPV DNA detection in physician-directed cervical specimens.

Methods:

Two pilots will be done, one at the Cleveland Clinic with the POI sampler and one at the University of Arizona using the Fournier device (with two different tip designs), in which we will recruit 150 consenting women attending a colposcopy clinic, including 50 women referred due to HSIL pap. Prior to undergoing a pelvic exam and insertion of the speculum, the attending physician will simulate self-collection of cervicovaginal specimens using, in alternating order, one of the new devices and a Dacron swab. After collection of the cervicovaginal specimens, women will then undergo a standard colposcopic evaluation but with an added cervical specimen collected from the os of the cervix to serve as the referent standard. Specimens (n=450, 3 paired specimens per woman, for the POI sampler pilot; n = 600, 4 paired specimens per woman, for the Fournier device pilot) will be tested in a masked fashion for oncogenic HPV DNA using Hybrid Capture 2 (HC2; Digene Corporation Gathersburg, MD) at the NCI HPV DNA core testing facility.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women age 21 and older

Non-pregnant, non-hysterectomized

EXCLUSION CRITERIA:

Pregnant women and women under the age of 21 will not be included in this study.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-01-09; Study Completion 2011-12-13

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Cleveland Clinical Health System, East Cleveland, Ohio

REFERENCES:
- [Background] Taylor LA, Sorensen SV, Ray NF, Halpern MT, Harper DM. Cost-effectiveness of the conventional papanicolaou test with a new adjunct to cytological screening for squamous cell carcinoma of the uterine cervix and its precursors. Arch Fam Med. 2000 Aug;9(8):713-21. doi: 10.1001/archfami.9.8.713. PMID 10927709
- [Background] Cramer DW. The role of cervical cytology in the declining morbidity and mortality of cervical cancer. Cancer. 1974 Dec;34(6):2018-27. doi: 10.1002/1097-0142(197412)34:63.0.co;2-b. No abstract available. PMID 4434331
- [Background] Fletcher A, Metaxas N, Grubb C, Chamberlain J. Four and a half year follow up of women with dyskaryotic cervical smears. BMJ. 1990 Sep 29;301(6753):641-4. doi: 10.1136/bmj.301.6753.641. PMID 2224218